CLINICAL TRIAL: NCT03478462
Title: An Open-Label, Dose Escalation, Efficacy, and Safety Study of CLR 131 in Children, Adolescents, and Young Adults With Select Solid Tumors, Lymphoma, and Malignant Brain Tumors
Brief Title: Dose Escalation Study of CLR 131 in Children, Adolescents, and Young Adults With Relapsed or Refractory Malignant Tumors Including But Not Limited to Neuroblastoma, Rhabdomyosarcoma, Ewings Sarcoma, and Osteosarcoma
Acronym: CLOVER-2
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cellectar Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCL-17-001
Record Dates: First submitted 2018-03-20; First posted 2018-03-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Solid Tumor; Pediatric Lymphoma; Pediatric Brain Tumor; DIPG; Neuroblastoma; Ewing Sarcoma; Rhabdomyosarcoma; Osteosarcoma
Keywords: medulloblastoma; ependymoma; high-grade glioma; glioblastoma; DIPG; diffuse-intrinsic pontine glioma; ATRT; atypical teratoid rhabdoid tumor; PNET; primitive neuroectodermal tumor; gliosarcoma; gliomatosis cerebri; neuroblastoma; rhabdomyosarcoma; Ewing sarcoma; osteosarcoma; DSRCT; desmoplastic small round cell tumor; sarcoma; malignant germ cell tumor; synovial sarcoma; rare cancer; Wilms tumor; lymphoma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma
MeSH Terms: conditions — Neuroblastoma; Sarcoma, Ewing; Rhabdomyosarcoma; Osteosarcoma; Medulloblastoma; Ependymoma; Glioma; Glioblastoma; Diffuse Intrinsic Pontine Glioma; Rhabdoid Tumor; Neuroectodermal Tumors, Primitive; Gliosarcoma; Neoplasms, Neuroepithelial; Desmoplastic Small Round Cell Tumor; Sarcoma; Sarcoma, Synovial; Wilms Tumor; Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — CLR1404

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CLR 131 (Experimental): CLR 131 intravenous administration
  Interventions: Drug: CLR 131

INTERVENTIONS:
Drug: CLR 131 — IV dose of CLR 131, increased/decreased by dose level; single or fractionated dose
  Other Names: I-131-CLR1404

SUMMARY:
The study evaluates CLR 131 in children, adolescents, and young adults with relapsed or refractory malignant solid tumors and lymphoma and recurrent or refractory malignant brain tumors for which there are no standard treatment options with curative potential.

DETAILED DESCRIPTION:
Even with standard, highly toxic multimodality therapies and salvage regimen, most pediatric patients with primary metastatic or relapsed solid tumors are confronted with a poor prognosis. For these patients there is currently no accepted successful treatment regimen. There is a need for new drugs, including targeted radiopharmaceuticals, preferably with cancer-specific uptake and broad applicability for these rare pediatric malignancies.

CLR 131 is a radioiodinated therapeutic that exploits the selective uptake and retention of phospholipid ethers (PLEs) by malignant cells. Cellectar Biosciences' novel cancer-targeted small-molecule compound (CLR1404) is radiolabeled with the isotope iodine-131 (I-131). CLR 131 has demonstrated tumor selective uptake across numerous adult and pediatric cancer cell types. Therapeutic efficacy has been demonstrated in various pediatric and adult-type cancer xenograft models, confirming the ability of CLR 131 to target tumors.

Based on the critical unmet medical need for effective agents with novel mechanisms of action in relapsed pediatric cancers and initial preclinical and clinical experience with radioiodinated CLR1404, Cellectar Biosciences has chosen to assess CLR 131 in a phase 1 pediatric trial.

ELIGIBILITY:
Inclusion Criteria:

All Patients

* Previously confirmed (histologically or cytologically) pediatric solid tumor (e.g., neuroblastoma, sarcoma), lymphoma (including Hodgkin's lymphoma), or malignant brain tumors that are clinically or radiographically suspected to be relapsed, refractory, or recurrent for which there are no standard treatment options with curative potential. Note: patients with diffuse intrinsic pontine glioma (DIPG) may enroll without histological or cytological confirmation.
* ≥ 2 years of age and ≤ 25 years of age at time of consent/assent
* If ≥ age 16 years, Karnofsky performance status of ≥ 60. If < age 16 years, Lansky performance status ≥ 60
* Platelets ≥ 75,000/µL (last transfusion, if any, must be at least 1 week prior to study registration, and, unless deemed medically necessary, no transfusions are allowed between registration and dosing)
* Absolute neutrophil count ≥ 750/µL
* Hemoglobin ≥ 8 g/dL (last transfusion must be at least 1 week prior to study registration, and, unless deemed medically necessary, no transfusions are allowed between registration and dosing)
* Using the bedside Schwartz formula, estimated GFR (creatinine clearance) > 60 ml/min/1.73m2
* Alanine aminotransferase < 3 × ULN
* Bilirubin < 2 × ULN
* Patients who have undergone autologous or allogeneic bone marrow transplant must be at least 3 months from transplant.
* Patients enrolling at total dose levels > 30 millicurie (mCi)/m2 must have availability or ability to collect an autologous hematopoietic stem cell back-up product prior to CLR 131 administration. At minimum, 2 x 10^6/kg cryopreserved CD34+ cells must be available.
* Patient or his or her legal representative is judged by the Investigator to have the initiative and means to be compliant with the protocol.

Patients with Pediatric Solid Tumor or Lymphoma

* At least 1 measurable lesion with longest diameter of at least 10 mm. Patients with a lesion(s) that are determined to be Metaiodobenzylguanidine (MIBG) or positron emission tomography (PET) positive may be enrolled at the investigator's discretion, even if not associated with a measurable lesion of at least 10 mm. Patients with neuroblastoma who have detectable disease may enroll provided they meet the requirements of the International Neuroblastoma Response Criteria.
* Patients with known brain metastases must have completed any radiotherapy or systemic treatments for brain metastases prior to enrollment; by investigator assessment be considered stable with no new signs or symptoms for at least 1 month, and on a stable dose of steroids (unchanged for three weeks prior to registration or on a steroid tapering regimen).

Patients with Recurrent or Refractory Brain Tumors

* At least 1 measurable lesion with longest diameter of at least 10 mm on any imaging sequence.
* Patients with previously known neurological deficits must be clinically stable at time of enrollment and able to complete all study related procedures. Patients with documented or newly diagnosed neurological deficits will be enrolled at the investigator's discretion.
* If patient receives steroids for neurological symptom control, the dose must be stable (unchanged for three weeks prior to registration) or on a steroid tapering regimen. Initiation of steroids per routine care immediately prior to CLR 131 dosing is acceptable.

Exclusion Criteria:

* Patients receiving active treatment for central nervous system metastases or those that are likely to require active treatment during anticipated participation in this trial. Patients with stable brain metastases treated with steroids may enroll at the investigator's discretion
* For solid tumor and lymphoma patients only, central nervous system involvement unless previously treated with surgery, systemic therapy, or radiotherapy with the patient neurologically stable. Patients with metastatic brain tumors that have been previously treated are allowed, provided the patient is neurologically stable (determined at the investigator's discretion).
* Antitumor therapy or investigational therapy, within 2 weeks of dosing. For certain types of radiation (craniospinal, total abdominal, whole lung [spot irradiation to skull-based metastases is not considered craniospinal radiation for the purposes of this study]), at least 3 months must have elapsed. No washout is required for palliative focal radiation. NOTE: Patients participating in non-interventional clinical trials (i.e., non-drug) are allowed to participate in this trial
* Patients previously treated with iodine-131 (131I)-MIBG who have already received a cumulative I-131 dose > 54 mCi/kg or who would exceed 54 mCi/kg by participating in this trial, are not eligible.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-04-30 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities (DLT) | up to 64 days
  DLT will be assessed by physical examination, vital signs, and laboratory values

SECONDARY OUTCOMES:
Identification of recommended phase 2 dose of CLR 131 in children, adolescents, and young adults | until non-tolerated dose is defined; dose escalation decision made upon review of data from a complete cohort (85 days after all subjects in cohort have received infusion)
  Dose and regimen to be used in Phase 2 trials of CLR 131 in children, adolescents, and young adults
Determination of preliminary antitumor activity of CLR 131 in children, adolescents, and young adults | through Day 85
  Response assessment per applicable criteria (e.g., Neuroblastoma Response Criteria (modified); RECIST 1.1; positron emission tomography response criteria in solid tumors (PERCIST); RANO)
Determination of therapeutic activity of CLR 131 in children, adolescents, and young adults | up to 22 days post initial infusion
  Assessment via 131-I/CLR 131 SPECT/CT scans
Determination of event free survival following CLR 131 infusion in children, adolescents, and young adults | 1 month to 5 years
  Time from first infusion of CLR 131 until progression or recurrence of disease
Determination of overall survival following CLR 131 infusion in children, adolescents, and young adults | 1 month to 5 years
  Time from first infusion of CLR 131 until death due to any reason
Determine dosimetry of CLR 131 in children, adolescents, and young adults | up to 15 days post initial infusion
  Assessment of dosimetry via whole body planar imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jarrod Longcor, Study Director — Cellectar Biosciences
Locations (8):
- United States (6):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Children's Hospital at Westmead, Westmead, New South Wales, Australia
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No